CLINICAL TRIAL: NCT05219214
Title: China Rheumatoid Arthritis Registry of Patients With Chinese Medicine
Acronym: CERTAIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Quan Jiang, MD, PhD, Professor, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Other Study IDs: Guang'anmen
Record Dates: First submitted 2022-01-01; First posted 2022-02-02 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chinese medicine group
  Interventions: Other: Chinese medicine

INTERVENTIONS:
Other: Chinese medicine — There are no restrictions on TCM therapy, including Chinese herbal medicine, Chinese patent medicine, external treatment, acupuncture and moxibustion, etc

SUMMARY:
A multi-center registration study of clinical characteristics of rheumatoid arthritis (RA) patients with Chinese medicine.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilled the rheumatoid arthritis classification criteria of 2010 American College of Rheumatology (ACR)/the European League Against Rheumatism (EULAR) .
* Aged 18 years and older.
* Be willing to accept CM therapies defined as Chinese herbal medicine, Chinese patent medicine, external treatment, acupuncture and moxibustion, etc

Exclusion Criteria:

* Refuse informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who meet the criteria will be enrolled from multi-centers in China.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Who Achieved Disease Activity Score for 28 Different Joints With C-reactive Protein Value (DAS28{CRP}) Remission (DAS28 <2.6) at Month 12 | Month 12
  DAS28 is a modification of the original DAS and is based on a count of 28 swollen and tender joints and is used to evaluate a participant's response to treatment. DAS 28 CRP utilizing joint scores from the following 28 joints: elbows, shoulders, elbow, wrists, metacarpal- phalangeal I-V, proximal interphalangeal I-V and knees and is calculated using the following formula: DAS28 (CRP) = 0.56*√(TJC28) +0.28*√(SJC28)+0.014*GH+0.36*ln(CRP+1)+0.96. Where TJC - Tender joint Count, SJC= Swollen Joint Count, (GH=participant assessment of disease activity using a 100 millimeter [mm] visual analogue scale with 0 = best, 100 = worst) and CRP= C reactive Protein (in [milligrams/liter] mg/L). It ranges between 0.96 and 8.61. High score (worse outcome) and low scores (better outcome).

SECONDARY OUTCOMES:
Change From Baseline in DAS28(CRP) at Month 12 | Baseline and month 12
  DAS28 is a modification of the original DAS and is based on a count of 28 swollen and tender joints and is used to evaluate a participant's response to treatment. DAS 28 CRP utilizing joint scores from the following 28 joints: elbows, shoulders, elbow, wrists, metacarpal- phalangeal I-V, proximal interphalangeal I-V and knees and is calculated using the following formula: DAS28 (CRP) = 0.56*√(TJC28) +0.28*√(SJC28)+0.014*GH+0.36*ln(CRP+1)+0.96. Where TJC-Tender joint Count, SJC= Swollen Joint Count, (GH=participant assessment of disease activity using a 100 millimeter [mm] visual analogue scale with 0 = best, 100 = worst) and CRP= C reactive Protein (in [milligrams/liter] mg/L). It ranges between 0.96 and 8.61. High score (worse outcome) and low scores (better outcome).Baseline was defined as the last available assessment prior to the start of study treatment. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Percentage of Participants Who Achieved Disease Activity Score for 28 Different Joints With erythrocyte sedimentation rate (DAS28{ESR}) Remission (DAS28 <2.6) at Month 12 | Month 12
  DAS28 is a modification of the original DAS and is based on a count of 28 swollen and tender joints and is used to evaluate a participant's response to treatment. DAS 28 ESR utilizing joint scores from the following 28 joints: elbows, shoulders, elbow, wrists, metacarpal- phalangeal I-V, proximal interphalangeal I-V and knees and is calculated using the following formula: DAS28 (ESR) = 0.56*√(TJC28) +0.28*√(SJC28)+0.014*GH+0.7*ln(ESR). Where TJC - Tender joint Count, SJC= Swollen Joint Count, (GH=participant assessment of disease activity using a 100 millimeter [mm] visual analogue scale with 0 = best, 100 = worst) and ESR= erythrocyte sedimentation rate (in millimeter/hour] mm/hr). . High score (worse outcome) and low scores (better outcome).
Change From Baseline in DAS28(ESR) at Month 12 | Baseline and month 12
  DAS28 is a modification of the original DAS and is based on a count of 28 swollen and tender joints and is used to evaluate a participant's response to treatment. DAS 28 ESR utilizing joint scores from the following 28 joints: elbows, shoulders, elbow, wrists, metacarpal- phalangeal I-V, proximal interphalangeal I-V and knees and is calculated using the following formula: DAS28 (ESR) = 0.56*√(TJC28) +0.28*√(SJC28)+0.014*GH+0.7*ln(ESR). Where TJC - Tender joint Count, SJC= Swollen Joint Count, (GH=participant assessment of disease activity using a 100 millimeter [mm] visual analogue scale with 0 = best, 100 = worst) and ESR= erythrocyte sedimentation rate (in millimeter/hour] mm/hr).. High score (worse outcome) and low scores (better outcome).Baseline was defined as the last available assessment prior to the start of study treatment. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Percentage of Participants Who Achieved DAS28(CRP) Remission (DAS28 <2.6) at All Time Points | through study completion, once every three months
  DAS28(CRP) remission is defined as a DAS28 score of <2.6 points. The DAS index combines information relating to the number of swollen and tender joints. The DAS28 is a modification of the original DAS and is based on a count of 28 swollen and tender joints and is used to evaluate a participant's response to treatment. DAS 28 CRP utilizing joint scores from the following 28 joints: elbows, shoulders, elbow, wrists, metacarpal- phalangeal I-V, proximal interphalangeal I-V and knees and is calculated using the following formula: DAS28 (CRP) = 0.56*√(TJC28) +0.28*√(SJC28)+0.014*GH+0.36*ln(CRP+1)+0.96. Where TJC - Tender joint Count, SJC= Swollen Joint Count, (GH=participant assessment of disease activity using a 100 mm visual analogue scale with 0 = best, 100 = worst) and CRP= C reactive Protein (in mg/L). It ranges between 0.96 and 8.61. High score (worse outcome) and low scores (better outcome).
Percentage of Participants Who Achieved DAS28(ESR) Remission (DAS28 <2.6) at All Time Points | through study completion, once every three months
  DAS28 is a modification of the original DAS and is based on a count of 28 swollen and tender joints and is used to evaluate a participant's response to treatment. DAS 28 ESR utilizing joint scores from the following 28 joints: elbows, shoulders, elbow, wrists, metacarpal- phalangeal I-V, proximal interphalangeal I-V and knees and is calculated using the following formula: DAS28 (ESR) = Joint Count, (GH=participant assessment of disease activity using a 100 millimeter [mm] visual analogue scale with 0 = best, 100 = worst) and ESR= erythrocyte sedimentation rate (in millimeter/hour] mm/hr). . High score (worse outcome) and low scores (better outcome).
Title:Change From Baseline in DAS28(CRP) at All Assessment Time Points | through study completion, once every three months
  DAS28 is a modification of the original DAS and is based on a count of 28 swollen and tender joints and is used to evaluate a participant's response to treatment. DAS 28 CRP utilizing joint scores from the following 28 joints: elbows, shoulders, elbow, wrists, metacarpal- phalangeal I-V, proximal interphalangeal I-V and knees and is calculated using the following formula: DAS28 (CRP) = 0.56*√(TJC28) +0.28*√(SJC28)+0.014*GH+0.36*ln(CRP+1)+0.96. Where TJC - Tender joint Count, SJC= Swollen Joint Count, (GH=participant assessment of disease activity using a 100 mm visual analogue scale with 0 = best, 100 = worst) and CRP= C reactive Protein (in mg/L). It ranges between 0.96 and 8.61. High score (worse outcome) and low scores (better outcome). Baseline was defined as the last available assessment prior to the start of study treatment. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline.
Title:Change From Baseline in DAS28(ESR) at All Assessment Time Points | through study completion, once every three months
  DAS28 is a modification of the original DAS and is based on a count of 28 swollen and tender joints and is used to evaluate a participant's response to treatment. DAS 28 ESR utilizing joint scores from the following 28 joints: elbows, shoulders, elbow, wrists, metacarpal- phalangeal I-V, proximal interphalangeal I-V and knees and is calculated using the following formula: DAS28 (ESR) = Joint Count, (GH=participant assessment of disease activity using a 100 millimeter [mm] visual analogue scale with 0 = best, 100 = worst) and ESR= erythrocyte sedimentation rate (in millimeter/hour] mm/hr). . High score (worse outcome) and low scores (better outcome). Baseline was defined as the last available assessment prior to the start of study treatment. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline.
Percentage of Participants With American College of Rheumatology's (ACR) 20/50/70 Response Rates at All Assessment Time Points | through study completion, once every three months
  DAS28(CRP) scores were categorized using EULAR response criteria. Response at a given time point was defined based on the combination of current DAS28 score and the improvement in the current DAS28 score relative to Baseline. The definition of no response, moderate response and good response was as follows: Current DAS28 <=3.2 and DAS28 decrease from Baseline (>1.2=good response), (>0.6 to <=1.2 = moderate response) and (<=0.6 =no response). Current DAS28 >3.2 to <=5.1 and DAS28 decrease from Baseline value (>1.2 =moderate response), (>0.6 to <=1.2 = moderate response) and (<=0.6 =no response). Current DAS28 >5.1 and DAS28 decrease from Baseline value (>1.2=moderate response), (>0.6 to <=1.2 = no response) and (<=0.6 =no response). If the post-Baseline DAS28(CRP) score was missing, then the corresponding EULAR category was set to missing.
Title:Percentage of Participants in Clinical Disease Activity Index (CDAI) Remission at All Assessment Time Points | through study completion, once every three months
  CDAI combines information relating to the number of swollen and tender joints, in addition to a measure of general health from both the participants and the physician. CDAI utilizing joint scores from the following 28 joints: elbows, shoulders, elbow, wrists, metacarpal- phalangeal I-V, proximal interphalangeal I-V and knees and is calculated using the following formula: CDAI =TJC28 + SJC28 + GH + GP Where TJC - Tender joint Count, SJC= Swollen Joint Count, (GH=participant assessment of disease activity and GP=physician assessment of disease activity using a 10 cm visual analogue scale with 0 = best, 100 = worst). It ranges between 0 and 76. High score indicates worse outcome, low score indicates better outcome. Remission was achieved for a non-missing CDAI value <=2.8.
Title:Percentage of Participants in Simple Disease Activity Index (SDAI) Remission at All Assessment Time Points | through study completion, once every three months
  SDAI combines information relating to the number of swollen and tender joints, in addition to a measure of general health from both the participants and the physician and acute phase reactants. The SDAI utilizing joint scores from the following 28 joints: elbows, shoulders, elbow, wrists, metacarpal-phalangeal I-V, proximal interphalangeal I-V and knees. It is calculated using the following formula: SDAI = TJC28 + SJC28 + GH + GP + CRP Where TJC - Tender joint Count, SJC= Swollen Joint Count, (GH=participant assessment, GP= physician assessment of disease activity using a 10 centimetre [cm] visual analogue scale [VAS] with 0 = best, 10 = worst), and CRP= C reactive Protein (in mg/L). It ranges between 0.1 and 86. High score indicates worse outcome, low score indicates better outcome. Baseline was defined as the last available assessment prior to the start of study treatment. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Change From Baseline in Chinese Patient-reported Activity Index with Rheumatoid Arthritis (CPRI-RA) at All Assessment Time Points | through study completion, once every three months
  CPRI-RA is the first rheumatoid arthritis Patient Reported Outcome(Pro) scale in China that has achieved expert consensus.The scale contains 11 items, including joint pain (item 1), swelling (item 2), morning stiffness (item 3), local skin temperature (item 4), upper limb activity function (item 5), lower limb activity function (item 6), fatigue (item 7), muscle soreness (item 8), appetite (Item 9) Irritability or anxiety (item 10) and difficulty in daily life (item 11). Each item is scored 0, 1, 2 and 3 respectively according to the four grades from none to there and from light to heavy, and then the total score is calculated according to the weight.Total score calculation formula = 1.43×(item 1) + 0.93×(item 2) + 0.40×(item 3)+1. 09×(item 4)+ 0.11×(item 5) + 0.18×(item 6) + 0.24×(item 7) + 0. 04×(item 8)+ 1.17 × (Item 9)+ 0. 19 ×(item 10) + 0. 02 ×(item 11). Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) at All Assessment Time Points | through study completion, once every three months
  HAQ-DI is 20-question instrument that assesses the degree of difficulty a person has in accomplishing tasks in eight functional areas;dressing and grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities. Each functional area contains at least two questions. For each question, there is a four level response set that is scored from 0 (without any difficulty) to 3 (unable to do). If aids or devices or physical assistance are used for a specific functional area and the maximum response of this functional area is 0 or 1 the according value is increased to a score of 2. HAQ-DI is only calculated if there are at least 6 functional area scores available. The average of these non-missing functional area scores defines the continuous HAQ-DI score ranging from 0 to 3. Baseline was defined as the last available assessment prior to the start of study treatment. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Participants' sharp score or modified total Sharp score(mTSS) score of wrist bone destruction at All Assessment Time Points | through study completion, once every three months
  Sharp evaluation is mainly a method to evaluate the bone destruction of wrist in patients with rheumatoid arthritis. The 27 parts of the hand and wrist were used as scoring points, and the scores were added from the two aspects of erosion score and narrowing degree of joint cavity: 0 for no bone erosion, 5 for extensive bone erosion and loss, and 2-4 between the two; 0 points for no stenosis, 1 point for local stenosis, 2 points for diffuse stenosis with an area of 50%, 3 points for diffuse stenosis with an area of > 50%, and 4 points for ankylosis.On this basis, van der heiide revised the mTSS to reduce the 27 scoring sites of the hand and wrist to 17 erosion evaluation sites and 18 joint cavity narrowing evaluation sites.
Number of Participants With Hematologic System Events at All Assessment Time Points | through study completion, once every three months
  The participants were tested with leucocyte count,platelet count,hemoglobin content and d-dimer test for regular metabolic function evaluation.The number of participants experiencing metabolic abnormal events have been reported.
Number of Participants With Metabolic Abnormal Events at All Assessment Time Points | through study completion, once every three months
  The participants were tested with blood lipid [total cholesterol(TC), triglyceride(TG), low density lipoprotein cholesterol(LDL-C)], blood glucose (Glu), liver and kidney function [aspartate aminotransferase(AST), alanine aminotransferase(ALT), gama-glutamyltransferase(GGT), Urea(Ur), Crea(Cr)] for regular metabolic function evaluation .The number of participants experiencing metabolic abnormal events have been reported.
Number of Participants With Cardiac Events | Up to 24 months
  Electrocardiograph(ECG) and ultrasonic cardiogram were used to evaluate cardiac function.Baseline was defined as the last available assessment prior to the start of study treatment. The number of participants experiencing Cardiac events have been reported.
Number of Participants With Pulmonary Events | Up to 24 months
  Pulmonary assessments were performed to determine the number of participants with pulmonary events including persistent cough, persistent dyspnea, and persistent Diffusing capacity of the lung for carbon monoxide (DLCO). Persistent is defined as any event with duration >=15 days. Baseline was defined as the last available assessment prior to the start of study treatment. The number of participants experiencing pulmonary events have been reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, China

REFERENCES:
- [Derived] Ma XL, Xia CM, Chang T, Liu ZX, Yang YC, Yao CH, Liu WX, Gong X, Jiang Q. Effectiveness and Safety of Biqi Capsules in 2,267 Patients with Rheumatoid Arthritis: A Real-World Clinical Study. Chin J Integr Med. 2026 Jan 15. doi: 10.1007/s11655-026-4137-5. Online ahead of print. PMID 41540164
- [Derived] Yao CH, Zhang C, Song MG, Xia CM, Chang T, Ma XL, Liu WX, Liu ZX, Liu JM, Tang XP, Liu Y, Liu J, Peng JY, He DY, Huang QC, Gao ML, Yu JP, Liu W, Zhang JY, Zhu YL, Hou XJ, Wang HD, Fang YF, Wang Y, Su Y, Tian XP, Lyu AP, Gong X, Jiang Q. Glucocorticoid Discontinuation in Patients with Rheumatoid Arthritis under Background of Chinese Medicine: Challenges and Potentials Coexist. Chin J Integr Med. 2025 Jul;31(7):581-589. doi: 10.1007/s11655-025-4212-3. Epub 2025 Jun 24. PMID 40553362
- [Derived] Gong X, Liu WX, Li D, Peng QW, Xia CM, Chang T, Guan JZ, Song MG, Zhang FY, Tang XP, Liu Y, Liu J, Peng JY, He DY, Huang QC, Gao ML, Yu JP, Liu W, Zhang JY, Zhu YL, Hou XJ, Wang HD, Fang YF, Wang Y, Su Y, Tian XP, Su X, Meng QL, Wen SY, Wang B, Li ZG, Liu J, Jiang H, Hu Y, Li HL, Wei SF, Zhu WH, Lyu AP, Zhang C, Jiang Q; CERTAIN Group. China rheumatoid arthritis registry of patients with Chinese medicine (CERTAIN): Rationale, design, and baseline characteristics of the first 11,764 enrollees. Phytomedicine. 2022 Sep;104:154236. doi: 10.1016/j.phymed.2022.154236. Epub 2022 Jun 14. PMID 35797864